CLINICAL TRIAL: NCT07182552
Title: Phase I Clinical Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics of NTB003 in Healthy Participants
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Chia-tai Tianqing Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTB003-101
Record Dates: First submitted 2025-08-18; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: TED

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NTB003 dose 1, dose 2, dose 3, dose 4 (Experimental)
  Interventions: Drug: NTB003
- Placebo dose 1, dose 2, dose 3, dose 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NTB003 — NTB003 dose 1, dose 2, dose 3, dose 4
  Arms: NTB003 dose 1, dose 2, dose 3, dose 4
Drug: Placebo — Placebo dose 1, dose 2, dose 3, dose 4
  Arms: Placebo dose 1, dose 2, dose 3, dose 4

SUMMARY:
This study is a randomized, double-blind, dose-escalation Phase I clinical trial to evaluate the safety, tolerability, and pharmacokinetic/pharmacodynamic characteristics of NTB003 injection in healthy volunteers.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, dose-escalation Phase I clinical trial to evaluate the safety, tolerability, and pharmacokinetic/pharmacodynamic characteristics of NTB003 injection in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ensure good communication with the Investigator, understand and comply with all requirements of the study, voluntarily participate in the trial, and sign the informed consent form.

  2. participants aged between 25 and 45 inclusive at the time of signing the informed consent form.

  3. Body mass index (BMI) is 19.0 kg/m2≤BMI≤26.0 kg/m2, and men must weigh ≥50 kg and women must weigh≥45 kg.

  4. Physical health and do not have any clinical diseases (including respiratory system, circulatory system, digestive system, nervous system, blood system, genitourinary system, endocrine system diseases) or mental illness (including depression, schizophrenia, etc.) during the screening interview.

  5. Physical examination, electrocardiogram, vital signs, laboratory and other related examinations are normal or abnormalities are of no clinical significance at screening.

  6. Agree to use reliable contraceptive methods with their partners during the trial; female volunteers of childbearing age must have a negative pregnancy test before the first use of the study drug.

Exclusion Criteria:

1. Known or suspected allergy to the investigational drug or any of its components, or predisposition to allergy.
2. Previous treatment with any anti-insulin-like growth factor-1 receptor (IGF-1R) monoclonal antibody.
3. Presence of scars, tattoos, moles, tenderness, bruising, erythema, induration, or damage at the intended injection site.
4. Difficulty with blood collection, inability to tolerate venous indwelling catheterization, or a history of syncope due to venipuncture.
5. Abnormal or did not have results for hepatitis B surface antigen, hepatitis C virus antibody, combined human immunodeficiency virus (HIV) antigen/antibody test, or Treponema pallidum antibody (TP-Ab).
6. History or suspected history of diabetes mellitus, or fasting blood glucose or glycated hemoglobin (HbA1c) above the upper limit of normal during screening.
7. History of ear diseases, ear surgery, hearing impairment, or a family history of hearing disorders.
8. History of thymic diseases such as thymoma or myasthenia gravis, or autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis, or inflammatory bowel disease.
9. Use of any medications within 2 weeks prior to screening, including prescription drugs, over-the-counter drugs, herbal medicines, traditional Chinese medicines, and dietary supplements.
10. Any active or suspected bacterial, viral, or fungal infection within 4 weeks prior to screening, such as common cold, viral syndrome, influenza-like symptoms.
11. Receipt of live attenuated or inactivated vaccines within 4 weeks prior to screening, or planned vaccination with such vaccines during the study period.
12. Underwent surgical procedures within 3 months prior to screening, or plans to undergo surgery during the study period.
13. Participation in any other clinical trial and receipt of an investigational drug within 3 months prior to screening.
14. Blood donation or significant blood loss (>400 mL), receipt of blood transfusion or blood products within 3 months prior to screening, or plans to donate blood or blood components during the study or within 3 months after completion.
15. Current smoker or history of smoking more than 5 cigarettes per day within 3 months prior to screening, or inability to abstain from tobacco products during the study.
16. History of alcohol abuse or regular alcohol consumption within 6 months prior to screening, defined as more than 14 units of alcohol per week (1 unit = 360 mL beer, 45 mL spirits with 40% alcohol, or 150 mL wine); unwillingness to abstain from alcohol or alcohol-containing products during the study; or abnormal/unperformed breath alcohol test results.
17. History of drug abuse or use of soft drugs (e.g., cannabis) or hard drugs (e.g., cocaine, phencyclidine) within 1 year prior to screening; or positive/unperformed urine drug screening results.
18. Special dietary requirements incompatible with a standardized diet.
19. Occurrence of acute illness during the screening phase or prior to study drug administration.
20. Any other condition that, in the opinion of the investigator, may interfere with the study or make the subject unsuitable for participation.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability, including the incidence of treatment-emergent adverse events (TEAEs), treatment-related TEAEs (TRAEs), and serious adverse events (SAEs) | Day 0 up to 154 days for healthy participants
  Safety and tolerability, including the incidence of treatment-emergent adverse events (TEAEs), treatment-related TEAEs (TRAEs), and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Pharmacokinetic parameter Cmax | Day 0 up to 154 days
Pharmacokinetic parameter Tmax | Day 0 up to 154 days
Pharmacokinetic parameter AUC | Day 0 up to 154 days
Pharmacokinetic parameter T1/2 | Day 0 up to 154 days
Incidence of anti-drug antibody (ADA) development in NTB003 treated participants over time | Day 0 up to 154 days
PD indicator IGF-1 concentration and changes relative to baseline | Day 0 up to 154 days

CONTACTS AND LOCATIONS:
Locations (1):
- Aerospace Center Hospital, Beijing, China